CLINICAL TRIAL: NCT00235404
Title: Specialized Treatment and Care Intervention at a Primary Level in a Nursing Home Compared to Conventional Treatment at a Hospital: a Randomized Controlled Trial.
Brief Title: Randomized Controlled Trial of Health Care to Elderly Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK 037-03
Record Dates: First submitted 2005-10-07; First posted 2005-10-10 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Congestive Heart Failure; Angina Pectoris; Asthma; Pneumonia; Fractures
Keywords: Treatment of elderly.; Nursing home.; Rehabilitation.; Readmissions.
MeSH Terms: conditions — Heart Failure; Angina Pectoris; Asthma; Pneumonia; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermediate community hospital (Experimental)
  Interventions: Other: Multicomponent treatment
- Usual care (Active Comparator)
  Interventions: Other: usual care

INTERVENTIONS:
Other: Multicomponent treatment — Specialized care in preparing recharge to home
  Arms: Intermediate community hospital
Other: usual care — Usual recharge directly from hospital to home
  Arms: Usual care

SUMMARY:
To study the efficacy of multicomponent treatment and care for patients with acute illness or deterioration of a chronic disease at a nursing home in primary health care compared to traditional treatment at hospital.

DETAILED DESCRIPTION:
Managers at St. Olavs University Hospital and the City of Trondheim local authority decided in 2001 to establish a reinforced department at a nursing home with a multicomponent approach to patient treatment.

In the study treatment at a nursing home will be compared with conventional treatment in ordinary hospital beds in medical, surgical and orthopedic departments at a hospital. Participating doctors at the hospital together with general practitioners shall develope inclusion criteria through Delphi technique. Eligible participants will be hospitalized from their ordinary home and expected to return to home after treatment. When an eligible patient is identified and accepted for inclusion, randomization will be performed by the Clinical Research Department at the Faculty of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Participating doctors at the hospital together with general practitioners shall develope inclusion criteria through Delphi technique.

Exclusion Criteria:

* Participating doctors at the hospital together with general practitioners shall develope exclusion criteria through Delphi technique.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2003-09; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Number of readmissions | Within 60 days
Number of deaths | Within 12 months
Need of home nursing services | within 12 months

SECONDARY OUTCOMES:
Costs | Within 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roar Johnsen, Study Chair — The Norwegian University of Science and Technology (NTNU)
Locations (1):
- Faculty of Medicine, The Norwegian University of Science and Technology (NTNU), Trondheim, Norway

REFERENCES:
- [Result] Garasen H, Windspoll R, Johnsen R. Intermediate care at a community hospital as an alternative to prolonged general hospital care for elderly patients: a randomised controlled trial. BMC Public Health. 2007 May 2;7:68. doi: 10.1186/1471-2458-7-68. PMID 17475006
- [Result] Garasen H, Magnussen J, Windspoll R, Johnsen R. [Elderly patients in hospital or in an intermediate nursing home department--cost analysis]. Tidsskr Nor Laegeforen. 2008 Jan 31;128(3):283-5. Norwegian. PMID 18264150
- [Result] Garasen H, Windspoll R, Johnsen R. Long-term patients' outcomes after intermediate care at a community hospital for elderly patients: 12-month follow-up of a randomized controlled trial. Scand J Public Health. 2008 Mar;36(2):197-204. doi: 10.1177/1403494808089685. PMID 18519285